CLINICAL TRIAL: NCT03650530
Title: The Family Talk Intervention Among Families With Childhood Cancer
Brief Title: The Family Talk Intervention in Pediatric Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Malin Lövgren, Assiciate Professor, Ersta Sköndal University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ErstaSUC
Record Dates: First submitted 2018-08-20; First posted 2018-08-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Oncology
Keywords: Family-centred intervention; Support program; The Family Talk Intervention

STUDY DESIGN:
Intervention Model Description: An intervention study with a single group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Family Talk Intervention (Experimental): These families will participate in a psychosocial support program.
  Interventions: Other: The Family Talk Intervention

INTERVENTIONS:
Other: The Family Talk Intervention — The family meets two interventionists at six time points.
  Other Names: Beardslee's Family Intervention

SUMMARY:
Even though most children with cancer now survive the ill child has to go through painful treatments which include suffering and uncertainty for all family members. The overall aim is to evaluate a modified version of the Family Talk Intervention (FTI) among families affected by childhood cancer. The goals of FTI are to increase family communication, the family members' resilience, knowledge about the illness, and thereby reduce the family members' long-term psychosocial well-being. Specific aims are to assess the feasibility (Aim 1) and the possible effects of the FTI (Aim 2).

Two to three months after diagnosis families at one of six pediatric oncology units in Sweden will be recruited to FTI. All families at this unit who have a child (with cancer and/or sibling) in the age of 6 to 19 will be asked to participate. The recruitment will continuing for 9 months.

The core elements in the intervention are to support: 1) the families in talking about the illness and related subjects, 2) the parents in understanding the needs of their children and how to support them, and 3) the families in identifying their strengths and how to use them. FTI entails six meetings with two interventionists (with the whole family and with the individual members of the family) at 1-2 weekly intervals.

Questionnaires, interviews and field notes will be used to evaluate the intervention. Time points for data collection: before the intervention starts (baseline), directly after the intervention (follow-up 1) and 6 months after baseline (follow-up 2).

Since few intervention studies (if any) of this kind have been carried out in pediatric oncology in Sweden to date, this study fills a knowledge gap. Research has described how cancer affects the whole family, and the importance of an open and honest communication about the illness in order to reduce the psychological suffering. The interventions presented here are likely to improve communication within the family, which may reduce the risk of long-term psychological distress for all family members.

DETAILED DESCRIPTION:
Previous research in pediatric oncology and evaluations from the Swedish Childhood Foundation, which focusing on parents', the ill child's, and the siblings' experiences, conclude that much remains to be done regarding support to families affected by childhood cancer. As there is no scientifically evaluated family-centered psychosocial intervention in pediatric oncology in Sweden intervention studies are needed. This present study, described below, fills a part of this knowledge gap. The overall aim is to evaluate a modified version of the Family Talk Intervention (FTI) among families affected by childhood cancer. The goals of FTI are to increase family communication, the family members' resilience, knowledge about the illness, and thereby reduce the family members' long-term psychosocial well-being. Specific aims are to assess the feasibility (Aim 1) and the possible effects of the FTI (Aim 2).

This is an intervention study that primarily focuses on feasibility. It will consist of an intervention group based on families affected by childhood cancer. One of the children in the family, the ill child or the sibling(s), have to be between 6-19 years old and the inclusion of families will be conducted approximately 2-3 months after the cancer diagnosis or relaps. The whole family or a part of the family can participate in the intervention. A minimum is that at least one adult and one child in the age 6-19 can participate. To participate, the family members have to understand and talk Swedish. All families that meet the inclusion criteria at the pediatric oncology unit at Astrid Lindgren Children's Hospital will be asked for participation from September 2018 to May 2019. Nurses at the clinic will identify the families that meet the inclusion criteria's. Information about the study will be sent home to the families by the researchers. One to two weeks later the interventionists will contact the families by phone, inform them about the study, and asked them about participation. Those who are willing to participate will be asked for informed consent.

FTI is a preventive method originally developed for families with a parent with an affective disorder who had children aged 6-18 years. The over-arching aims of the method are not traditional psychotherapeutic intervention. They are instead to support an open, honest and child-centered family communication, and increase understanding of the disease. The intervention also aims to promote parental awareness concerning protective factors (as well as identification of such), such as well-functioning school life, relationships and hobbies among their children. Even if the intervention was developed for families with a parent with depression it has also been tested among families with a severely ill parent who has young children, with positive results. The core elements in the intervention are to: 1) support the families in talking about the illness and related subjects 2) support the parents in understanding the needs of their children and how to support them, and, 3) support the families in identifying their strengths and how to use them. One of the most important principles is respect for the parents. It is important to emphasize the parents' expertise regarding their children.

Since pediatric oncology is yet another context, the intervention has been slightly modified by the research group together with individuals who educate persons in FTI in Sweden. The modified FTI entails six meetings at 1-2 weekly intervals with five extra meetings. The interventionists, who work in pairs, are educated in FTI and have clinical experiences of working with families affected by seriously illness (e.g. as a nurse, counselor, etc.). To support the interventionists a supervisor/educator in FTI will be available. The FTI is manual-based and the interventionists are following a special protocol (here called the logbook). The meetings with the families are held at a place chosen by the families.

Meetings 1-2: include only the parent(s) and focus on the parents' experiences of their situation as well as the consequences of the cancer diagnosis for each family member. During the meeting, each child's situation will be discussed including strengths, problems, worries, the situation in school and with friends, and their social network. The knowledge of the disease will also be a focus. The parent(s) will formulate the goal of the intervention. They can also formulate questions that the interventionist(s) will ask the children in meetings 3.

Meeting 3: interviews will be held with each child (without the parents) concerning the child's life situation, feelings, understanding of the disease, questions and hobbies. The relationship with their parents is discussed as well as the child's social network. The interventionist(s) identifies protective factors from the child's narrative (e.g. well-functioning school life and relationships with friends) as well as risk factors (e.g. poor social network). The child can also formulate questions for the parents and what he/she wants to discuss during the family meeting.

Meeting 4: includes the parent(s) and focuses on the planning of the family meetings. The child's thoughts and questions serve as a guide for the upcoming family meeting.

Meeting 5: is preferably led by the parent(s) to facilitate ongoing and continuous communication within the family, and consists of questions and issues raised earlier by each family member. This family meeting can be seen as a starting point for communication within the family.

Meeting 6: is a follow-up with all family members, held preferably within a month of meeting 5. The meeting is guided by the family members' needs, e.g. communication and parenting.

Various strategies will be implemented during the different meetings including conversation technique, books and different techniques of expression such as drawing and writing. For example the interventionist(s) will use mapping of the children's social network as one technique to assess the support that children receive.

In case of that the intervention not can be finished due to special circumstances extra meetings will be available (meeting 7-11).

Mixed methods, i.e. questionnaires, interviews and notes, will be used to evaluate the FTI.

The primary focus for this study is on the feasibility (Aim 1). Interviews and notes from the logbooks will be analyzed with content analysis and the study process will be observed. As this is a first study in this context, the results of the potential effects (Aim 2) will indicate the direction for further studies. The potential effects will be explored with descriptive statistics (data from the questionnaires) focusing on within effects where descriptive trends of e.g. family communication will be explored. However, the main part of Aim 1 will be answered by interview data from the families, the interventionist and by observations. This study will also contribute to a power calculation for a larger study in this context.

ELIGIBILITY:
Inclusion Criteria:

* One of the children in the family, the ill child or the sibling(s), have to be between 6-19 years old
* At least one adult and one child in the age 6-19 from the same family have to participate
* The family members have to understand and talk Swedish

Exclusion Criteria:

* Families with children only under 6 years or over 19 years
* Families were only the parent(s) or the children want to participate
* Families that do not speak and write Swedish.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Survey data on family communication | Baseline (before the intervention start), follow-up 1 (after the end of the intervention, approximately 2 months after baseline) and follow-up 2 (approximately 6 months after baseline)
  Changed family Communication will be measured with the Family Communication Scale. The minimum possible score is 10 points, and the maximum possible score is 50 points. A higher score indicates a better level of family communication. Total score of 10-29 represent very low level of communication, 30-35 low level of communication, 36-39 moderate level of communication, 40-44 high level of communication and 45-50 very high level of communication. A step within the framework of very high/high/moderate/low/very low represents a change. Study-specific questions will also be used.

SECONDARY OUTCOMES:
Survey data on psychosocial health | Baseline (before the intervention start), follow-up 1 (after the end of the intervention, approximately 2 months after baseline) and follow-up 2 (approximately 6 months after baseline)
  For the children: Changed psychosocial wellbeing using the Pediatric Quality of Life Inventory version 4.0. To create the Psychosocial Health Summary Score, the mean is computed as the sum of the items over the number of items answered in the Emotional, Social, and School Functioning Scales. A 4.5 change in PedsQL score for Child self-report has been determined as a minimum Clinical meaningful difference.
Survey data regarding knowledge about the illness | Baseline (before the intervention start), follow-up 1 (after the end of the intervention, approximately 2 months after baseline) and follow-up 2 (approximately 6 months after baseline)
  Changed knowledge about the illness: Study specific questions will be used, for example open-ended questions to children about the namn of the illness, if someone has talked to them about the treatment, the prognosis, etc.
Survey data on family satisfaction | Baseline (before the intervention start), follow-up 1 (after the end of the intervention, approximately 2 months after baseline) and follow-up 2 (approximately 6 months after baseline)
  Changed family satisfaction measured by the Family Satisfaction Scale. The sum of all items represents a total score ranged 10-50. Total score of 10-29 represent very low satisfaction, 30-35 low satisfaction, 36-39 moderate satisfaction, 40-44 high satisfaction and 45-50 very high satisfaction. A step within the framework of very high/high/moderate/low/very low represents a change.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Lövgren, PhD, Principal Investigator — Ersta Sköndal Bräcke University College
Locations (1):
- Ersta Sköndal Bräcke University College, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD is not planed to be shared with other researchers outside the group.

REFERENCES:
- [Derived] Eklund R, Lovgren M. The Family Talk Intervention in Pediatric Oncology: Ill Children's Descriptions of Feasibility and Potential Effects. J Pediatr Hematol Oncol Nurs. 2022 May-Jun;39(3):143-154. doi: 10.1177/27527530221068423. Epub 2022 Feb 17. PMID 35467434
- [Derived] Iveus K, Eklund R, Kreicbergs U, Lovgren M. Family bonding as a result of the family talk intervention in pediatric oncology: Siblings' experiences. Pediatr Blood Cancer. 2022 Mar;69(3):e29517. doi: 10.1002/pbc.29517. Epub 2021 Dec 31. PMID 34971075
- [Derived] Lovgren M, Kreicbergs U, Udo C. Family talk intervention in paediatric oncology: a pilot study protocol. BMJ Paediatr Open. 2019 Jan 31;3(1):e000417. doi: 10.1136/bmjpo-2018-000417. eCollection 2019. PMID 30815590